CLINICAL TRIAL: NCT05082493
Title: A Phase 1, Multicenter, Open-label, Dose Escalation Study of the Safety and Pharmacokinetics of Intravenously Infused Berubicin in Pediatric Patients With Progressive, Refractory, or Recurrent High Grade Gliomas
Brief Title: A Multicenter, Study of the Safety and Pharmacokinetics of Intravenously Infused Berubicin in Pediatric Patients With Progressive, Refractory, or Recurrent High Grade Gliomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: WPD Pharmaceuticals Sp. z o.o. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPD-201P
Record Dates: First submitted 2021-09-22; First posted 2021-10-19 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, multicenter, open-label, dose escalation study of intravenous Berubicin in pediatric patients. The purpose of this first-in-pediatrics study is to examine the safety, tolerability, and PK of Berubicin and to estimate its MTD and/or RP2D when administered to pediatric patients with progressive, refractory, or recurrent HGG who have completed at least 1 standard line of therapy. This study will also make a preliminary assessment of the antitumor activity of Berubicin in this patient population. An exploratory evaluation of quality of life will also be performed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Berubicin HCL - MTD phase (Experimental): Berubicin will be administered as 1-hour infusions each day for 3 consecutive days followed by 18 days off drug (ie, 21-day cycles). The starting dose is based on population PK modeling of data from adult studies and will be 1.20 mg/m2 (Dose Level 1). During the study, PK data will be incorporated into a PK model on an ongoing basis and may be used to inform dose escalation decisions
  Interventions: Drug: Berubicin Hydrochloride

INTERVENTIONS:
Drug: Berubicin Hydrochloride — Berubicin will be administered as 1-hour infusions each day for 3 consecutive days followed by 18 days off drug (ie, 21-day cycles). The starting dose is based on population PK modeling of data from adult studies and will be 1.20 mg/m2 (Dose Level 1). During the study, PK data will be incorporated into a PK model on an ongoing basis and may be used to inform dose escalation decisions

SUMMARY:
This is a Phase 1, multicenter, open-label, dose escalation study of intravenous Berubicin in pediatric patients. The purpose of this first-in-pediatrics study is to examine the safety, tolerability, and PK of Berubicin and to estimate its MTD and/or RP2D when administered to pediatric patients with progressive, refractory, or recurrent HGG who have completed at least 1 standard line of therapy. This study will also make a preliminary assessment of the antitumor activity of Berubicin in this patient population. An exploratory evaluation of quality of life will also be performed

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, dose escalation study of intravenous Berubicin in pediatric patients. The purpose of this first-in-pediatrics study is to examine the safety, tolerability, and PK of Berubicin and to estimate its MTD and/or RP2D when administered to pediatric patients with progressive, refractory, or recurrent HGG who have completed at least 1 standard line of therapy. This study will also make a preliminary assessment of the antitumor activity of Berubicin in this patient population. An exploratory evaluation of quality of life will also be performed.

This open-label, nonrandomized study is composed of a series of Dose Escalation Cohorts followed by an Expansion Cohort. The Dose Escalation Cohorts will utilize a standard "rules based" 3+3 design. A safety review committee (SRC) composed of, at a minimum, the principal investigators, the medical monitor(s), the sponsor's responsible medical officer (s), and an external expert in pediatric oncology will review all available study data at regular intervals and will make recommendations to the sponsor regarding dose escalations. Patients enrolled in the Expansion Cohort will be administered the MTD or RP2D identified during dose escalation. Safety, PK, efficacy, and quality of life evaluations will be performed for all patients throughout the study.

Berubicin will be administered as 1-hour infusions each day for 3 consecutive days followed by 18 days off drug (ie, 21-day cycles). The starting dose is based on population PK modeling of data from adult studies and will be 1.20 mg/m2 (Dose Level 1). During the study, PK data will be incorporated into a PK model on an ongoing basis and may be used to inform dose escalation decisions.

Dose Escalation and Stopping Rules: The Dose Escalation Cohorts will utilize a standard 3+3 design to determine an MTD and/or RP2D. All available information, including safety, PK, and efficacy, will be taken into account when making decisions regarding dose escalation. The 3 + 3 dose escalation procedures will be based on the following:

Enroll 3 patients initially. If no dose-limiting toxicities (DLTs; as defined in Safety Outcome Measures) occur, escalate dose to next dose level cohort.

If 1 patient out of 3 experiences a DLT, expand cohort up to 6 patients. If 1 patient out of 6 experiences a DLT, escalate to next dose level cohort. If ≥2 patients out of 6 experience a DLT, the MTD will have been exceeded; stop dose escalation, and review the next lower dose cohort. This may require enrollment of a further 3 patients if only 3 were dosed at a previous dose level.

Note that patients who experience a DLT may not necessarily be required to discontinue from the study, based on the judgement of the investigator. Patients who discontinue from a Dose Escalation Cohort before the end of the DLT evaluation period for reasons other than a DLT will be replaced.

Once the MTD or RP2D has been established, an Expansion Cohort will be initiated. Patients enrolled in the Expansion Cohort will receive the MTD or RP2D identified during Dose Escalation.

Patients may continue to receive additional cycles of Berubicin in the absence of clinical and/or neurologic deterioration or unacceptable toxicity as long as both the patient's legally authorized representative (LAR) and investigator agree that further therapy is in the patient's best interest. Patients with radiographic evidence of progression but who are clinically stable and are not experiencing significant neurologic decline (based on investigator assessments and Neurological Assessment in Neuro-Oncology [NANO] criteria) may remain on the study at the discretion of the investigator.

Patients will return for a follow-up assessment on Day 28, approximately 25 days after the last dose of Berubicin.

All patients, including those who discontinue study treatment for any reason, will continue to be followed (Post-Study Follow up) for further anti-tumor treatment and survival every 3 months until death, loss to follow-up, withdrawal of consent, or end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent of the patient's LAR, and assent when appropriate based on the patient's age and institutional guidelines, prior to any study-related procedure.

  2. Patients must have progressive, refractory, or recurrent HGG (WHO Grade III or IV).

  3. Age ≥2 to <18 years at the time of the first Berubicin dose. 4. Performance status score ≥50 (Lansky for research patients aged ≤16 years and Karnofsky for patients ˃16 years). Patients who are unable to walk because of paralysis but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.

  5. Patients must have completed at least 1 line of prior therapy. 6. Before the projected start of scheduled study treatment, the following time periods must have elapsed:
  1. 5 half-lives from any investigational agent.
  2. 4 weeks from cytotoxic therapy (except 23 days from temozolomide and 6 weeks from nitrosoureas).
  3. 6 weeks from antibody therapies.
  4. 4 weeks (or 5 half-lives, whichever is shorter) from other antitumor therapies.
  5. Patients who have received radiation therapy must be ≥6 weeks post the completion of local palliative radiation therapy (re-irradiation for progressive disease or upfront radiation therapy at initial diagnosis).

     7. Adequate organ function defined as:

  a. Bone marrow: i. Peripheral absolute neutrophil count ≥1000/mm3 ii. Hemoglobin ≥8 g/dL (may have received packed red blood cell transfusion) iii. Platelet count ≥100,000/mm3 (transfusion-independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) b. Renal function: i. Creatinine clearance or radioisotope glomerular filtration rate ≥70 mL/min/1.73 m2 or normal serum creatinine based on age c. Hepatic function: i. Total bilirubin (sum of conjugated + unconjugated) ≤1.5 × the upper limit of normal (ULN) for the institution ii. Alanine aminotransferase ≤3 × ULN for the institution iii. Serum albumin ≥2 g/dL d. Neurologic function: i. Patients with seizure disorder may be enrolled if the seizure disorder is well controlled, as determined by the investigator.

  e. Cardiac function (left ventricular ejection fraction [LVEF]): i. Fractional shortening ≥27% or LVEF ≥50% by echocardiogram or multigated radionuclide study (MUGA) 8. All adverse events (AEs) Grade >1 related to prior therapies (chemotherapy, radiation therapy, and/or surgery) must be resolved to Grade 1 or baseline level, except for alopecia and sensory neuropathy Grade ≤2 or other Grade ≤2 AEs not constituting a safety risk based on the investigator's judgment.

  9. For postpubertal patients: Female patients must agree to use highly effective contraception during the period of the study and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use highly effective contraception during the period of the study and for at least 3,5 months (no less than 104 days) after completion of treatment. Details are provided in the full protocol.

  10. Female patients of childbearing potential aged 10 years or older must have a negative serum or urine pregnancy test.

  11. MRI of the brain and entire spine (including all sites of disease), within 10 days prior to start of study drug.

  12. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the baseline MRI scan.

Exclusion Criteria:

* 1. Evidence of diffuse leptomeningeal disease or evidence of cerebrospinal fluid (CSF) dissemination.

  2. Known additional malignancy that is progressing or has required active treatment within 3 years of start of study drug.

  3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Berubicin or its excipients.

  4. Patients with any clinically significant, unrelated systemic illness (eg, significant pulmonary, hepatic [including Gilbert's syndrome], or other organ dysfunction) or psychiatric illness/social situations that would compromise the patient's ability to tolerate the study drug or study procedures or would likely interfere with the study procedures or results.

  5. Any known clinically significant active bacterial, fungal, or viral infection including hepatitis B or hepatitis C, or any underlying disease in the recent past that could compromise enrollment and the safety of the patient.

  6. Patient with a history of clinically significant, uncontrolled heart disease and/or repolarization abnormalities as documented by a standard 12 lead electrocardiogram (ECG).

  7. Known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias, or bradycardia, unless arrhythmia is controlled and after a cardiology consultation has cleared the patient to receive Berubicin. Patients receiving therapeutic agents known to prolong QT interval will be excluded; however, the use of ondansetron is permitted. Patients with a history of congestive heart failure, myocardial infarction, or stroke in the last 3 months will be excluded.

  8. Congenital long QT syndrome or QTc >460 ms. 9. Patients receiving any other anticancer or investigational drug therapy. 10. Prior treatment with bevacizumab. 11. Current or planned participation in a study of another investigational agent or using an investigational device.

  12. Requirement for cytochrome P450 3A4 (CYP3A4)-inducing or inhibiting agents, with the exception of corticosteroids.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
• Dose Escalation Cohorts first outcome | 6 months
  To estimate the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of single-agent Berubicin administered after at least 1 prior line of therapy in pediatric patients with progressive, refractory, or recurrent HGG.
  To completely document the assessment of response, the measurements of the longest tumor dimension, and its perpendicular, of all target lesions should be recorded for the baseline and all subsequent follow-up exams. Changes in nontarget lesions and newly occurring lesions should also be described. The same method of assessment and the same technique should be used at baseline and during follow-up.
• Dose Escalation Cohorts second outcome | 6 months
  To estimate the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of single-agent Berubicin administered after at least 1 prior line of therapy in pediatric patients with progressive, refractory, or recurrent HGG.
  Tumor response criteria are determined by changes in size using the longest tumor dimension and its perpendicular. If multiple measurable lesions are present, a minimum of the 2 largest lesions should be measured; a maximum of 5 should be selected as target lesions. Target lesions should be selected on the basis of size and suitability for accurate repeated measurements. All other lesions will be followed as nontarget lesions. Only solid components of cystic/necrotic tumors should be measured.
• Expansion Cohort first outcome | 6 months
  To evaluate the safety of Berubicin administered at the MTD or RP2D to pediatric patients with progressive, refractory, or recurrent HGG who have completed at least 1 prior line of therapy The MTD is empirically defined as the highest dose level at which 6 patients have been treated with at most 1 patient experiencing a DLT and the next higher dose level has been determined to be not tolerated (≥2 out of 6 patients experience a DLT). The MTD estimation will be limited to evaluable patients and toxicity assessments from the first cycle of Berubicin treatment (21 days).
• Expansion Cohort second outcome | 6 months
  To evaluate the safety of Berubicin administered at the MTD or RP2D to pediatric patients with progressive, refractory, or recurrent HGG who have completed at least 1 prior line of therapy The RP2D is a multifactorial endpoint that considers toxicity as well as additional determinants (eg, efficacy, pharmacodynamics) to define the optimal Phase 2 dose on the basis of available clinical safety and efficacy data. It is usually a dose in which there is ≤20% dose-limiting toxicity; however, it can be further defined by exploration of doses that maximize efficacy in the presence of minimal safety concerns.

IPD SHARING:
Plan to Share IPD: No